CLINICAL TRIAL: NCT03463018
Title: A Phase 2 Randomized, Double-Blind, Parallel-Group, Placebo Controlled Fixed-Dose Study of Echinacea Angustifoliae Root Extract (AnxioCalm) in Healthy Subjects With Subthreshold Symptoms of Anxiety
Brief Title: Echinacea Angustifolia (AnxioCalm) in Anxiety
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment error; Inclusion criteria not met
Sponsor: EuroPharma, Inc. (Industry)
Collaborators: Simon Khechinashvili University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EP-1003; EP-02-2017 (Other: Sponsor)
Record Dates: First submitted 2018-03-02; First posted 2018-03-13 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Generalized Anxiety Disorder
Keywords: Echinacea, Subthreshold Anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Echinacea extract

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Echinacea angustifolia (Experimental): 20 mg tablet of Echinacea angustifolia root extract standardized for a specific alkamide profile, two tablets twice daily (total daily dose of 80 mg) for two weeks
  Interventions: Dietary Supplement: Echinacea angustifolia
- Placebo (Placebo Comparator): Identical excipients as in the experimental arm, without the active ingredient
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Echinacea angustifolia — 20 mg tablet of Echinacea angustifolia, standardized for echinacoside (not less than 3%) and alkamides (not less than 0.8%)
  Arms: Echinacea angustifolia
Dietary Supplement: Placebo — Placebo tablet containing matching excipients to the active intervention
  Arms: Placebo

SUMMARY:
This study evaluates whether Echinacea angustifolia (AnxioCalm) is a safe and effective treatment for mild to moderate Generalized Anxiety Disorder (GAD) symptoms. Half the participants will receive Echinacea angustifolia and half will receive placebo.

DETAILED DESCRIPTION:
Echinacea angustifolia root extract (AnxioCalm), standardized for the content of echinacoside and its alkamide profile, is intended to be used for 'amelioration of sub-threshold and mild anxiety which are risk factors in the development of Generalized Anxiety Disorder (GAD) and depression' in symptomatic people 'who are not eligible for anxiolytic medication.' Existing medical interventions, which require long periods of repeated administration, have significant safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age (all races and ethnicity)
* Meet Diagnostic and Statistical Manual of Mental Disorders (DSM IV) any criteria for Generalized Anxiety Disorder (GAD from 5 to 9)
* mild to moderate symptom severity on the Beck Anxiety Inventory (BAI from 8 to 15)
* Hamilton Anxiety Rating Scale (HAM-A) score from 14 to 17
* Hospital Anxiety and Depression Scale (HADS-A) [hospital anxiety and depression scale - anxiety subscale] - 8-10
* Participants score 45-57 points of above on either the state or trait anxiety subscale of the State and Trait Anxiety Inventory of Speilberger (STAI)
* Able to understand and provide signed informed consent
* Able to participate in a 5-week study

Exclusion Criteria:

* Any diagnosed DSM-IV Axis II disorder
* Current DSM IV Axis I diagnosis of Major Depressive Disorder in the 6 month that precede the study. [to exclude confounding psychiatric factors]
* Danger of suicidality
* Treatment with Echinacea preparations in the 3 month that precede the study
* Psychotropic medication (especially anxiolytics) in the 3 month that precede the study
* Psychotherapy in the 3 month that precede the study
* Allergic reactions to plants of the Asteraceae family (Echinacea species, etc.)
* Treatment for AIDS or cancer
* Pregnant or lactating women
* Unstable medical condition (e.g., hypothyroidism, hypertension, myocardial infarction within 1 month, neoplastic condition)
* Alcohol or drug dependence within 3 months
* Allergy to Echinacea preparation
* Allergy to plants of the Asteraceae family (e.g., ragweed, asters, chrysanthemum)
* Allergy to mugwort, radioallergosorbent test (RAST), or birch tree pollen Concurrent tranquilizer, antidepressant or mood stabilizer therapy;
* Subjects receiving anti-anxiety medication (e.g., benzodiazepine, venlafaxine, buspirone, or SSRI)
* Concurrent use of over-the-counter anti-anxiety and/or antidepressant preparations (e.g., chamomile, St. John's Wort, Kava kava)
* Women of child-bearing potential not willing to employ a medically proven form of contraception (e.g., condoms, oral contraceptives, etc)
* Any other condition that precludes participation according to the judgement of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating (HAM-A) | 14 days
  The Hamilton Anxiety Rating Scale (HAM-A) is a physician rating scale consisting of 14 items measuring psychic and somatic anxiety. Each item is scored on a scale of 0 (none) to 4 (severe) where a total score of 14-17 = Mild Anxiety, 18-24 = Moderate Anxiety, 25-30 = Severe Anxiety. The primary outcome is the change over time in the baseline HAM-A score rating for AnxioCalm versus placebo.
State-Trait Anxiety Inventory (STAI) | 14 days
  The State-Trait Anxiety Inventory (Form Y, 6 item) is a six item patient rating scale consisting of anxiety present and anxiety absent items. Each item is rated from 1 (not at all) to 4 (very much). For scoring, positive items (calm, relaxed, content) are reverse scored [1=4, 2=3, 3=2, 4=1], the six scores are totaled, and multiplied by 20/6. A normal score is approximately 34-36.The primary outcome is the change over time in the baseline STAI score for AnxioCalm versus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Janelidze, PhD MD, Principal Investigator — Simon Khechinashvili University Hospital, I.Chavchavadze 33, 0162, Tbilisi, Georgia
Locations (1):
- Simon Skechinashvili University Hospital, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No